CLINICAL TRIAL: NCT04369560
Title: Virtual Histology of the Bladder Wall for Bladder Cancer Staging; A Novel Intravesical Contrast-Enhanced MRI for Bladder Cancer Staging
Brief Title: Virtual Histology of the Bladder Wall for Bladder Cancer Staging
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jodi Maranchie (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Jodi Maranchie, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HCC 20-054
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Urinary Bladder Neoplasms
Keywords: TURBT; Complete Cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Magnetic Resonance Imaging; Ferrosoferric Oxide

STUDY DESIGN:
Intervention Model Description: Diagnostic Test - Magnetic Resonance Imaging
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Magnetic Resonance Imaging (Experimental): Prior to planned surgical resection, subjects will undergo a single Magnetic Resonance Imaging study: a single breath-hold pre-contrast image followed by sterile placement of a temporary urethral catheter for instillation of a 50mL solution containing Gadobutrol (4 mM) plus ferumoxytol (5 mM) and a second, single breath hold post-contrast image.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Drug: Gadobutrol intravesical administration (4mM); Drug: Ferumoxytol intravesical administration (5 mM)

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — 60-cm wide bore 3T scanner (Siemens AG, Erlangen, Germany) with a 32-channel pelvic phased-array coil placed over the bladder.
Drug: Gadobutrol intravesical administration (4mM) — A paramagnetic macrocyclic gadolinium-based contrast agent administered intravenously for use in magnetic resonance imaging. Contrast-enhancement is a result of the neutral complex of gadolinium and dihydroxy-hydroxymethylpropyl- tetraazacyclododecane-triacetic acid (butrol).
  Other Names: Image result for other names for Gadobutrol Gadavist
Drug: Ferumoxytol intravesical administration (5 mM) — An iron preparation (Fe3O4) approved for intravenous treatment of anemia in the setting of renal failure, comprised of superparamagnetic iron oxide nanoparticles which are coated by a semi-synthetic carbohydrate shell in an isotonic, neutral pH solution.
  Other Names: FERAHEME

SUMMARY:
This is a phase Ib study of the safety and performance of a novel intravesical contrast-enhanced Magnetic Resonance Imaging protocol for determination of bladder cancer stage prior to transurethral resection of bladder tumor (21 subjects) or prior to radical cystectomy for muscle invasive disease (21 subjects). Subjects will undergo a single MRI study: a pre-contrast, single breath hold image followed by sterile placement of a temporary urethral catheter for instillation of a 50mL solution containing Gadobutrol (4 mM) plus ferumoxytol (5 mM) and then a second, post-contrast image. Images will be reviewed by two dedicated abdominal radiologists, who are blinded to the pathologic staging, for determination of tumor presence and depth of bladder wall penetration.

DETAILED DESCRIPTION:
Twenty one patients with at least one cystoscopically confirmed papillary bladder tumor, who have been scheduled for Transurethral Resection of Bladder Tumor (TURBT) for surgical extirpation and staging, and twenty-one patients with histologically confirmed, muscle invasive transitional cell carcinoma of the bladder who have been scheduled for definitive radical cystectomy with curative intent will be recruited for a single study Magnetic Resonance Imaging to be performed between 1 and 6 days prior to their scheduled procedure.

Magnetic Resonance Imaging of all the enrolled patients will be performed on a 60-cm, wide-bore, 3T scanner (Siemens AG, Erlangen, Germany) with a 32-channel pelvic phased-array coil placed over the bladder using radial k-space sampling technique for volumetric free breathing acquisition with NCM enhanced StarVIBE57. Un-enhanced fast spoiled gradient-echo images with fat suppression will be obtained prior aseptic instillation of 50cc of a novel contrast mixture (NCM) of Gadobutrol (4 mM) plus Ferumoxytol (5 mM) in sterile water through a temporary urethral catheter. The catheter will then be removed and the patient repositioned in the scanner to obtain post-contrast images. All the image datasets will be linearly registered to the subject to ensure that regions of interest represent the same anatomical location at all time points. Post-contrast T1, pre-contrast T1 and deltaT1 will be measured from the acquired images. Two radiologists blinded to the pathologic findings will evaluate the Magnetic Resonance images to assign a radiologic tumor stage that will be compared with the subsequent pathologic stage determined at time of surgery. Following the MRI study, subjects will proceed with their surgical procedure as scheduled per standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 90 years of age
2. Able to understand and willing to sign a written informed consent document
3. A papillary tumor identified by cystoscopy that has been scheduled for TURBT OR histologically proven MIBC that is clinically localized and amenable to surgical resection with curative intent.
4. Performance status of ECOG 0 or 1
5. Normal renal function as defined as creatinine less than 1.5 x institutional upper limit of normal (ULN) OR creatinine clearance greater than or equal to 50 mL/min/1.73 m2 by Cockcroft-Gault formula for subjects with creatinine levels greater than or equal to 1.5 x ULN.

Exclusion Criteria:

1. Severe hypersensitivity reaction to gadobutrol or ferumoxytol.
2. Severe claustrophobia that will prevent completion of the MRI study.
3. Any MRI-non-compatible implanted device, prosthetic or pacemaker.
4. Known or suspected metastatic disease.
5. Women with active pregnancy, lactation or plans to conceive
6. Untreated urinary tract infection
7. Known urethral stricture disease that would prohibit placement of foley catheter.
8. Any other conditions considered as unacceptable risk by the treating physician

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Magnetic Resonance Imaging assessment of depth of bladder wall penetration to predict pathologic stage determined at tumor resection | 4 weeks
  The assessment of clinical tumor stage assigned by the radiologist will be compared to the stage reported by the clinical pathologist following tumor resection to determine the overall accuracy of MRI for bladder cancer staging.

SECONDARY OUTCOMES:
Accuracy of Magnetic Resonance Imaging to detect residual/recurrent bladder tumor | 4 weeks
  Patients are typically scheduled for radical cystectomy after initial TURBT with or without neoadjuvant chemotherapy. MRI findings of bladder tumor will be compared with the areas of tumor identified on whole mount sectioning of the bladder to estimate the sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) of MRI for bladder cancer. Receiver operating characteristic (ROC) curve analysis will be used to estimate the tumor size threshold value for the diagnosis with MRI.
Rate of Adverse Events | 2 years
  Characterize the safety profile of MRI imaging following direct bladder instillation of a mixture of Gadobutrol and Ferumoxytrol (50mL in sterile water) via urethral catheter by soliciting and recording adverse events while on study.

CONTACTS AND LOCATIONS:
Overall Officials: Jodi K Maranchie, MD, Principal Investigator — Associate Professor
Locations (1):
- UPMC Hillman Cancer Center - Dept of Urology, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
1. What data will be shared? The investigators will share the accuracy of the MRI staging versus the traditional pathological staging.
  2. Who will have access to the data? The investigators and future researchers who provide the proper MTA, IRB, etc. will have access to the de-identified data.
  3. Where will the data to be shared be located? De-identified data will be kept on the UPMC cloud.
  4. When will the data be shared? The data will be available to share after final analysis and publication of results.
  5. How will researchers locate and access the data? A link to the Cloud folder will be provided.